CLINICAL TRIAL: NCT04229108
Title: A Feasibility Study Into a Self-recorded, Digital, Timed Up and Go Test Using the Medopad Platform for the General Public
Brief Title: Digitisation of the Timed Up and Go Test for the General Public
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Andrew Gvozdanovic (Industry)
Responsible Party: Sponsor-Investigator, Andrew Gvozdanovic, Clinical Manager, Medopad
Organization: Medopad (Industry)
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MEDOPAD007
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Medopad application
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Other): Will record traditional timed up and go followed by two digitised versions
  Interventions: Device: Medopad

INTERVENTIONS:
Device: Medopad — Timed up and go module of Medopad application. About page explains how to perform test and conditions, subsequent page contains timer, once completed test, commence on final page which has a number of short questions to complete

SUMMARY:
The question this feasibility study aims to answer is whether or not participants are able to accurately and reliably perform and self record the timed up and go test in a non-clinical environment using the Medopad application. This forms part of a larger question of whether or not a more frequently performed TUG test, could act as a physical activity marker.

DETAILED DESCRIPTION:
This is a single centre study which will take place in a mock clinical and non-clinical environment. The site-specific requirements including a clear space in which the participant can walk for 3m, and a firm chair with sturdy arms. The individuals performing the clinically led test must have experience in performing clinical examinations and be able to explain the steps involved in the Timed Up and Go in a clear and cohesive manner as judged by the study operators.

Participants will initially be asked to perform a clinician led 'Timed Up and Go' (TUG), this result will be recorded including:

1. Number of attempts
2. Use of arm rests to aid
3. Whether mobility aid is used

Each participant will be given a rest period of at least 10 minutes. Participants will be asked to download the Medopad application onto their own mobile device. Once onboarded, they will be shown how to use the TUG module and then asked to complete a non-clinician led TUG, this result will be digitally stored on the application. Participants will be instructed to carry out the TUG in the following manner: sit in an upright chair with arm rests, with no extra cushions or pillows on the seat. They will be advised to ideally use a firm chair of height ~46cm with arm rests. Whilst at home, they will be asked to place the 3m ruler down in front of the chair they plan to use, open up the application and enter the TUG module. At this point, they will be prompted to take a picture of their chair, they will then need to sit down and rest for 5 minutes and re-read through the TUG module information. After 5 minutes they will need to press the 'Go' button on the application and perform the test, pressing the 'Stop' button on completion.

Following this initial test, participants will then be asked to repeat this TUG in a week's time. They will be provided with a standardised 3 metre measuring device to ensure correct distance at home. After completion of the final TUG test, they will be asked to complete a short feedback questionnaire regarding their experience.

At each test performance, the participant will be asked to place a second mobile device with the Medopad application loaded. The motion capture module of this device's application with be initiated as the start of the test and record accelerometer and gyroscope data during the test's performance. It will then be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* English speaking
* Able to follow instructions and commands
* Assistance of 0 (but can use mobility aids)
* Low falls risk (no falls within the past year)
* Able and willing to perform at least 2 consecutive timed up and go tasks in a clinical setting, with at least a further repeat of the TUG task independently at home
* Ownership of an iOS or Android capable smartphone which can run the Medopad app

Exclusion Criteria:

* Cognitive disorders/impairment (MMSE ≤ 24) unless test to be performed by carer who feels this is appropriate
* Severe visual impairment (interfering with their ability to use the application)
* Physical impairment preventing safe use of the TUG test in the home environment
* Those without the appropriate facilities to perform the TUG at home (i.e no appropriate chair meeting minimum criteria)
* Unable to physically use the Medopad application
* Pregnancy
* Inability to consent to study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-27 (Estimated); Primary Completion 2020-02-06 (Estimated); Study Completion 2020-02-06 (Estimated)

PRIMARY OUTCOMES:
Time difference between traditional and digitised timed up and go test | 1-2 month
  The primary outcome measure will be to record the time taken to complete the traditional timed up and go test versus the time taken when the test is performed by non-clinicians in a non-clinical setting using the Medopad application TUG module. Time will be measured in minutes and seconds.

SECONDARY OUTCOMES:
Accelerometer data produced during the performance of all timed up and go tests. | 1-2 month
  Accelerometer data using a second mobile device in the patient's right pocket. Data will be measured in metres per second^2 in the x, y, and z axis of the phone.
Gyroscope data produced during the performance of all timed up and go tests. | 1-2 months
  Collect gyroscope data using a second mobile device in the patient's right pocket. This will measure angular velocity in degrees per second or revolutions per second.

OTHER OUTCOMES:
Qualitative research questionnaire into patient satisfaction with the study and timed up and go module | 1-2 month
  A questionnaire will be used to collect quantitative scaled data (1-5, with 1 being a worse outcome i.e least satisfied, least happy and 5 being associated with a better outcome, i.e more satisfied, most happy) surrounding: how satisfied participants were with the study process, how happy participants were with visual appearance of the application, and how happy participants were using the application. The questionnaire will also collect qualitative data on whether participants would be happy to use the digitised form of the TUG in the future (yes or no) and any areas to improve the study or application (free text).

IPD SHARING:
Plan to Share IPD: Undecided